CLINICAL TRIAL: NCT01697332
Title: Functional Applications of Hyperpolarized 129Xe MRI
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Funding ended prior to resolution of all equipment (polarizer) issues.
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Samuel Patz, Scientific Director, Center for Pulmonary Functional Imaging, Brigham and Women's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2012P001947; 5R01HL096471-04 (NIH)
Record Dates: First submitted 2012-09-26; First posted 2012-10-02 (Estimated); Results first posted 2018-04-17 (Actual); Last update posted 2018-04-17 (Actual); Status verified 2018-03

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Subjects with and without COPD (Experimental): All subjects will inhale hyperpolarized 129Xe gas and then have a MRI scan performed to measure lung function.
  Interventions: Drug: Hyperpolarized 129Xe gas

INTERVENTIONS:
Drug: Hyperpolarized 129Xe gas — 800cc of a gas mixture containing 129Xe and nitrogen will be inhaled by a subject. The subject will hold their breath for no more than 16 seconds while a MRI scan is performed. The gas mixture can contain between 20 and 100% xenon.

SUMMARY:
The overall objectives of our study are to determine the capabilities of hyperpolarized 129Xe MRI to measure lung function and its potential to sensitively detect pulmonary disease and its progression in COPD. We hypothesize that measurement of alveolar surface area, septal thickness, and capillary transit time measured with hyperpolarized 129Xe will correlate better with quality of life measures in COPD subjects than traditional diagnostic measures such as spirometry and Computed Tomography.

ELIGIBILITY:
Inclusion Criteria:

* Age 20-75

For Healthy nonsmoker subjects:

* No current physician diagnosed medical disease requiring active medication
* No smoking history, defined as less than 100 cigarettes smoked in a lifetime
* Normal spirometry: FEV1/FVC ≥ 0.70, FEV1 ≥ 80% predicted

For Subjects who have participated in the COPDGene Study

* Post-bronchodilator spirometry: FEV1 > 40% predicted

Exclusion Criteria:

* MR contraindications: e.g., electrical implants such as cardiac pacemakers, ferromagnetic implants such as prostheses, claustrophobia
* Pregnancy or suspected pregnancy
* Use of continuous oxygen
* Use of antibiotics and/or systemic corticosteroids (new prescription or increased dose) for an exacerbation of lung disease or any lung infection in the past four weeks
* Uncontrolled cancer, as defined as ongoing radiation therapy, ongoing chemotherapy
* A heart attack in the past three months

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2013-01 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Patz, PhD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham & Women's Hospital, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Subjects With and Without COPD
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Subjects With and Without COPD
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 1
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Baseline Statistics of Healthy Subjects
Description: Hyperpolarized 129Xe MRI scans will be performed on healthy subjects and the uptake of 129Xe in the pulmonary septal tissue will be measured as a function of time. From this data, the mean and distribution of three pulmonary functional parameters will be determined. The three measures are alveolar surface area per unit volume, septal thickness and capillary transit time through the gas exchange region.
Time Frame: 4 years
Population: No data collected or analyzed for this outcome measure.
Arm/Group | Subjects With and Without COPD
Number analyzed (Participants) | 0

2. Primary Outcome: Differences Between Healthy and Diseased COPD Subjects.
Description: Hyperpolarized 129Xe MRI measures of disease severity in GOLD Stage 1-3 subjects are more highly correlated with physical disabilities associated with their pulmonary disease than traditional tests of pulmonary function.
Time Frame: 4 years
Population: No data analyzed or collected for this outcome measure.
Arm/Group | Subjects With and Without COPD
Number analyzed (Participants) | 0

3. Primary Outcome: Spatial Heterogeneity
Description: Determine the degree to which the spatial heterogeneity of regional 129Xe measurements of pulmonary function in a single individual correlates with physical manifestations of disease severity. We hypothesize that measures of spatial heterogeneity will correlate highly with physical disability.
Time Frame: 4 years
Population: No data analyzed or collected for this outcome measure.
Arm/Group | Subjects With and Without COPD
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 4 years.
Arm/Group | Subjects With and Without COPD
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No